CLINICAL TRIAL: NCT04673006
Title: Risk of Bacterial Exposure to the Anesthesiologist's Face During Intubation and Extubation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0529
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Anesthesiologists Who Perform Endotracheal Intubation and Extubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — face shield swab culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anesthesiologists who will perform endotracheal intubation and extubation for general anesthesia: All anesthesiologists in this study will use face shield for facial protection. Face shield swab will be done before and after the procedures (intubation and extubation)

SUMMARY:
The practice of intubation and extubation is not without risks to the anesthesiologists. Especially, the face of health care worker is the body part most commonly contaminated by splashes and sprays of body fluids. The aim of this study is to determine the incidence of unrecognized exposure to the anesthesiologists' face during endotracheal intubation and extubation. We will perform face shield swab before and after the endotracheal intubation and extubation. All swabs will be cultured for 48 hours and the number of colony forming units before and after the procedures (intubation/extubation) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* anesthesiologists who perform endotracheal intubation and extubation for patients scheduled for endotracheal intubation for elective surgeries

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All anesthesiologists who perform endotracheal intubation and extubation will be included in this study. This study will be done only in patients who are scheduled for endotracheal intubation for elective surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Bacterial growth of face shield swab after the endotracheal extubation | Bacterial swab will be performed 5 minutes after the endotracheal extubation (after the confirmation of sufficient spontaneous breathing)
  All swab will be cultured for 48 hours and will be reported as no growth or by number of colony forming unit(CFU)s. The number of CFU of post-extubation swab will be compared with that of pre-extubation swab.

SECONDARY OUTCOMES:
Bacterial growth of face shield swab after the endotracheal intubation | Bacterial swab will be performed 5 minutes after the endotracheal extubation (after the confirmation of adequate mechanical ventilation)
  All swab will be cultured for 48 hours and will be reported as no growth or by number of colony forming unit(CFU)s. The number of CFU of post-intubation swab will be compared with that of pre-intubation swab.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, Principal Investigator — Severance Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No